CLINICAL TRIAL: NCT05181137
Title: A Phase 3 Study to Evaluate the Efficacy and Long-term Safety of SHR0302 Therapy in Subjects With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Phase 3 Study to Investigate the Efficacy and Safety of SHR0302 With Moderately to Severely Active Ulcerative Colitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSJ10135
Record Dates: First submitted 2021-12-10; First posted 2022-01-06 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ivarmacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 Active Experimental: SHR0302 Dose#1 (Experimental): SHR0302 Oral tablets taken once daily (QD) for 8 weeks SHR0302 Oral tablets taken once daily (QD)
  Interventions: Drug: SHR0302
- Part 1 Placebo Comparator: Placebo (Placebo Comparator): Placebo Oral tablets taken once daily (QD) for 8 weeks
  Interventions: Drug: Placebo
- Part 2 Active Experimental: SHR0302 Dose#2 (Experimental): SHR0302 Oral tablets taken once daily (QD) for 44 weeks
  Interventions: Drug: SHR0302
- Part 2 Placebo Comparator: Placebo (Placebo Comparator): Placebo Comparator: Maintenance Treatment Placebo Comparator: Placebo
  Interventions: Drug: Placebo
- Part 3 Active Experimental: SHR0302 Dose#2 (Experimental): SHR0302 Oral tablets taken once daily (QD) for 26 weeks
  Interventions: Drug: SHR0302

INTERVENTIONS:
Drug: SHR0302 — Oral tablets taken once daily (QD)
  Arms: Part 1 Active Experimental: SHR0302 Dose#1; Part 2 Active Experimental: SHR0302 Dose#2; Part 3 Active Experimental: SHR0302 Dose#2
Drug: Placebo — Oral tablets taken once daily (QD)
  Arms: Part 1 Placebo Comparator: Placebo; Part 2 Placebo Comparator: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multicenter Phase 3 study that will enroll approximately 368 subjects aged 18 to 75 years old with Moderately to Severely Active Ulcerative Colitis.

DETAILED DESCRIPTION:
This study consists of a screening period followed by a placebo-controlled Part 1 phase and then a placebo-controlled Part 2 phase. An open label Part 3 phase is open to subjects who: complete the Part 2, are considered non-responders following the Part 1, or have disease worsening during Part 2.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Part 1

1. Male or female subjects must be at least at ≥18 and ≤75 years of age
2. Subject has at least a three-month history of Ulcerative Colitis diagnosis at baseline.
3. Subject has active Ulcerative Colitis with a 9-point modified Mayo score of ≥ 5 at baseline, with an endoscopic subscore of ≥ 2
4. Subject is deemed by the physician as having inadequate response, loss of response or intolerance to at least one conventional treatment (oral 5-ASA, immunosuppressants or corticosteroids), or was previously exposed to anti-TNF therapy (e.g., infliximab, adalimumab) or other biological treatment (e.g., vedolizumab) having

Discontinued the treatment for:

* Infliximab: a minimum of 8 weeks prior to baseline.
* Adalimumab: a minimum of 10 weeks prior to baseline.
* Ustekinumab: a minimum of 14 weeks prior to baseline.
* Vedolizumab: a minimum of 17 weeks prior to baseline.

Inclusion Criteria for Part 2 1. Subject has completed Part 1 and achieved clinical response at week 8

Inclusion Criteria for Part 3

1. Subject has completed the 8-week Part 1 and was classified as not meeting clinical response criteria. OR Subject has discontinued treatment early in the Maintenance phase due to disease worsening OR Subject has completed the Maintenance phase.

Study Exclusion Criteria for Part 1

Exclusion Criteria:

1. Subject has a diagnosis of indeterminate colitis, or clinical findings suggestive of Crohn'sDisease.
2. Subject with Ulcerative Colitis, which is confined to a proctitis (distal 15 cm or less).
3. Treatment naïve subject diagnosed with Ulcerative Colitis (without previous exposure to any of the following therapies for UC treatment: oral 5-ASA, corticosteroids, immunosuppressants, or biological treatments).
4. Subject is displaying clinical signs of ischemic colitis, fulminant colitis or toxic megacolon.
5. Subject had previous surgery as a treatment for Ulcerative Colitis or likely to require surgery during the study period.
6. Subject has evidence of pathogenic bowel infection. Subjects had Clostridium difficile or other intestinal infection within 30 days of screening endoscopy or test positive at screening for C.difficile toxin or other intestinal pathogens.
7. Subject currently has or has a history of active tuberculosis (TB) or latent TB infection.
8. Subject is receiving any of the following therapies:

   * Azathioprine/6-mercaptopurine, methotrexate, thalidomide within 7 days prior to baseline.
   * Cyclosporine, mycophenolate, tacrolimus within 4 weeks prior to baseline.
   * Interferon therapy within 8 weeks prior to baseline.
   * Intravenous corticosteroids or rectally administered formulation of corticosteroids or 5- ASA within 2 weeks prior to baseline.
9. Subject had any prior treatment with lymphocyte-depleting agents/therapies (such as CamPath® [alemtuzumab], alkylating agents [e.g., cyclophosphamide or chlorambucil], total lymphoid irradiation, etc.). Subjects who have received rituximab or other selective B lymphocyte depleting agents are eligible if they have not received such therapy for at least 1 year prior to baseline.
10. Subject has previously received JAK inhibitors, such as tofacitinib, baricitinib, upadacitinib, filgotinib.
11. Subject with evidence of clinically relevant laboratory abnormalities which may affect subject safety or interpretation of study results at screening
12. Subject has a screening 12-lead ECG that demonstrates clinically relevant abnormalities
13. Subject currently has or had:

    * A clinically significant infection within 1 month of baseline (e.g., those requiring hospitalization or parenteral antimicrobial therapy or have opportunistic infections).
    * A history of more than one episode of herpes zoster, or disseminated zoster (single episode).
    * Any infection otherwise judged by the investigator to have the potential for exacerbation by participation in the study.
    * Any infection requiring antimicrobial therapy within 2 weeks of screening.
14. Subject has current immunization with any live virus vaccine or history of immunization with any live virus vaccine within 8 weeks of baseline.
15. Subject with a first-degree relative with a hereditary immunodeficiency.
16. Subject with a history of any lymphoproliferative disorder (such as EBV-related lymphoproliferative disorder, as reported in some subjects on other immunosuppressive drugs), history of lymphoma, leukemia, multiple myeloma, or signs and symptoms that are suggestive of current lymphatic disease.
17. Subject has any condition possibly affecting oral drug absorption e.g., gastrectomy, or clinically significant diabetic gastroenteropathy, or certain types of bariatric surgery such as gastric bypass. (Procedures such as gastric banding, gastric balloon that simply divide stomach into separate chambers, are NOT exclusionary.) Subject has undergone significant trauma or major surgery within 4 weeks of baseline.
18. Women who are pregnant or lactating, or planning pregnancy while enrolled in the study. Male who plan to donate sperm during the study and within 30 days after the last dose of study drug.
19. Subject who has a history of alcohol or drug abuse with less than 6 months of abstinence prior to baseline that in the opinion of the investigator will preclude participation in the study.
20. Subject with malignancies or with a history of malignancies with exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin.
21. Subject infected with human immunodeficiency virus (HIV) or hepatitis B or C viruses.
22. Subject has received any investigational drug or device within 3 months, or 5 half-lives (if known) prior to baseline.
23. Subject is receiving or expected to receive prohibited concomitant medication(s) in the 4 weeks prior to the first dose of study drug and through follow-up visit.
24. Any other condition which in the opinion of the investigator would make the subject unsuitable for inclusion in the study.
25. Subject with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, urogenital, nervous system, musculoskeletal, skin, sensory, endocrine (including uncontrolled diabetes or thyroid disease), or hematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the Investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
26. Subject with a history of thromboembolic events, including deep vein thromboses (DVT), pulmonary embolism (PE), and those with known inherited conditions that predispose to hypercoagulability.

Study Exclusion Criteria for Parts 2 and 3

1. Subject with any clinically significant condition at the end of 8-week Induction treatment from Part 1 Induction phase, and Part 2 Maintenance Phase that in the opinion of investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis.
2. Subject who, in the opinion of the investigator or sponsor, is unlikely to be cooperative or able to comply with study procedures, or any other condition which in the opinion of the investigator would make the subject unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2021-11-05 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical remission at week 8 (Part 1) | 8 weeks
  The percentage of subjects in clinical remission at week 8.
Clinical remission at week 52 (Part 2) | 52 weeks
  The percentage of subjects in clinical remission at week 52.

SECONDARY OUTCOMES:
Endoscopic remission at week 8 (Part 1) | 8 weeks
  The percentage of subjects with endoscopic remission at week 8.
Clinical response at week 8 (Part 1) | 8 weeks
  The percentage of subjects with clinical response at week 8.
Change from baseline in partial Mayo score at week 2, 4, and 8 (Part 1) | 8 weeks
  Change from baseline in partial Mayo score at week 2, 4, and 8.
Change in total Mayo score and 9-point modified Mayo score at week 8 (Part 1) | 8 weeks
  Change in total Mayo score and 9-point modified Mayo score at week 8.
Subjects with endoscopic remission (Part 2) | 52 weeks
  The percentage of subjects with endoscopic remission at week 52.
Subjects with clinical response at week 52 (Part 2) | 52 weeks
  The percentage of subjects with clinical response at week 52.
Change from baseline in partial Mayo score at week 12, 16, 24, 32, 40, and 52 (Part 2) | 52 weeks
  Change from baseline in partial Mayo score at week 12, 16, 24, 32, 40, and 52.
Change in total Mayo score and 9-point modified Mayo score at week 52 (Part 2) | 52 weeks
  Change in total Mayo score and 9-point modified Mayo score at week 52.
Subjects in corticosteroid-free remission at week 52 (Part 2) | 52 weeks
  Percentage of subjects in corticosteroid-free remission at week 52.
Subjects who maintain clinical remission at week 52 (Part 2) | 52 weeks
  Percentage of subjects who maintain clinical remission at week 52
Subjects in clinical remission per partial Mayo score at week E26 (Part 3) | 26 weeks (extension)
  The percentage of subjects in clinical remission per partial Mayo score at week E26.
Subjects in corticosteroid-free remission per Partial Mayo score at week E26 (Part 3) | 26 weeks (extension)
  The percentage of subjects in corticosteroid-free remission per Partial Mayo score at week E26.
Change from baseline in Partial Mayo score at week E2, E12, and E26 (Part 3) | 26 weeks (extension)
  Change from baseline in Partial Mayo score at week E2, E12, and E26.

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Chen, Study Director — Reistone Pharma
Locations (113):
- United States (23):
  - Digestive Health Specialists, Dothan, Alabama
  - Om Research LLC, Lancaster, California
  - Yale University, New Haven, Connecticut
  - IHS Health, Kissimmee, Florida
  - Dade Research Center, Miami, Florida
  - Gastro Florida, Pinellas Park, Florida
  - One Health Research Clinic Atlanta, LLC, Norcross, Georgia
  - John Hopkins University, Columbia, Maryland
  - Michigan Medical, Ann Arbor, Michigan
  - Research Institute of Michigan, Chesterfield, Michigan
  - NY Scientific, Brooklyn, New York
  - DiGiovanna Institute for Medical Education & Research, North Massapequa, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Charlotte Gastroenterology & Hepatology P.L.L.C, Charlotte, North Carolina
  - DDSI, Oklahoma City, Oklahoma
  - Central Sooner Research, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Omni Clinical Research, Houston, Texas
  - UTMB Health, League City, Texas
  - University of Utah, Salt Lake City, Utah
  - McGuire Research Institute, Richmond, Virginia
  - IACT Health, Suffolk, Virginia
  - Advocate Aurora Health - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- China (59):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Military Area General Hospital/Seventh Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Tsinghua University Changgung Hospital, Beijing, Beijing Municipality
  - Army Medical Center of PLA, Chongqing, Chongqing Municipality
  - Chongqing People's Hospital, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospitial of Xiamen University, Xiamen, Fujian
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science and Technoloy, Luoyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Hena
  - Jingzhou First People's Hospital, Jingzhou, Hubei
  - Affiliated Taihe Hospital of Hubei University of Medicine, Shiyan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Huai'an First People's Hospital, Huai'an, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing General Hospital of Nanjing Military Command, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Subei People's Hospital of Jiangsu province, Yangzhou, Jiangsu
  - Shengjing Hospital Of China Medical University, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Longhua Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Shanxi, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Tianjin medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Union Medical Center, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University of Traditional Chinese Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jinhua Municipal Central Hospical, Jinhua, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Georgia (4):
  - Curatio, Jsc, Tbilisi
  - JSC Infectious Diseases, AIDS and Clinical Immunology Research Center, Tbilisi
  - LTD Central University Clinic After Academic N. Kipshidze, Tbilisi
  - LTD The First Medical Center, Tbilisi
- Poland (13):
  - CLINSANTE Clinical Research Centre Ewa Galczak-Nowak, Malgorzata Trzaska, Bydgoszcz
  - MZ BADANIA Slowik Zymla General Partnership, Knurów
  - "Landa" Specialist Doctor's Offices, Krakow
  - PLEJADY Medical Centre, Krakow
  - AMED Medical Centre Branch in Lodz, Lodz
  - Oswiecim Clinical Trial Centre, Oświęcim
  - Private Healthcare Institution Specialist Clinics Termedica, Poznan
  - Dariusz Kleczkowski Specialist Medical Practice, Sopot
  - Torun Gastrology Centre "Gastromed", Torun
  - MDM Healthcare Centre, Warsaw
  - WIP Warsaw IBD Point, Warsaw
  - Medical Centre Oporow, Wroclaw
  - ETG Zamosc, Zamość
- Ukraine (14):
  - Communal Nonprofit Enterprise "Cherkasy Regional Hospital of Cherkasy Oblast Council", Cherkasy
  - Regional Municipal Non-commercial Enterprise "Chernivtsi Emergency Medical Hospital", Chernivtsi
  - Public Non-Profit Enterprise "Regional Clinical Hospital under Ivano-Frankivsk Regional Council", Ivano-Frankivsk
  - Public Non-Profit Institution: O.O. Shalimov City Clinical Hospital #2 under Kharkiv City Council, Kharkiv
  - Public Non-Profit Enterprise "Khmelnytskyi Regional Hospital" under Khmelnytskyi Regional Council, Khmelnytskyi
  - Clinical Hospital "Feofaniia", Kyiv
  - Medical Center "Consylium Medical", Kyiv
  - Medical Center OK!Clinic+ of the Company with Limited Liability International Institute of Clinical Research, Kyiv
  - Municipal Enterprise "Volyn Regional Clinical Hospital" of Volyn Regional Council, Lutsk
  - Communal Noncommercial Enterprise of Lviv Regional Council "Lviv Regional Clinical Hospital", Lviv
  - Public Non-Profit Enterprise under Sumy Regional Council "Sumy Regional Clinical Hospital", Sumy
  - Communal Non-Commercial Enterprise: Vinnytsia City Clinical Hospital #1, Vinnytsia
  - Public Non-Profit Enterprise "City Hospital #6" under Zaporizhia City Council, Zaporizhia
  - "Medibor Plus" Llc, Zhytomyr

IPD SHARING:
Plan to Share IPD: No